CLINICAL TRIAL: NCT02002481
Title: Vergleich Der Qualität Der Kardiopulmonalen Reanimation Durch Professioneller Helfer (Notärzte / Rettungsassistenten) während Lufttransporten
Brief Title: Comparison of the Quality of CPR by Professional Helpers (Emergency Physicians / Paramedics) During Flights
Acronym: flights
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Dr. med. Stefan Braunecker, Anesthesiologist, Researcher, University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-289
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): 10 minutes ALS-CPR in a normal environment
- Transport (Experimental): 10 minutes ALS-CPR during a transport
  Interventions: Other: transport

INTERVENTIONS:
Other: transport — The manikin will be resuscitated during a transport in a vessel by a professional team (emergency physician / paramedic).
  Arms: Transport

SUMMARY:
Investigation of the influence of narrowness and unusual circumstances on the CPR-quality

DETAILED DESCRIPTION:
Even for paramedics and emergency physicians, the resuscitation of patients with cardiac arrest remains a challenge. Previous studies have shown that the cardiac output varies widely even under normal ambient conditions. Especially the mean frequenices of cardiac compression varies from 60 to 160/min, as well as the now-flow-time. Aim of this study is to investigate how narrowness and movement during a transport affect the CPR-performance.

For this, we examine the impact of the common transport options (air and ground) on the outcome-varity on a manikin. The subjects for this study are professional rescuers (emergency physicians / paramedics) who perform a 10 minute ALS-CPR in either normal circumstances (resuscitation-room) or during transportation.

ELIGIBILITY:
Inclusion Criteria:

* emergency physician
* paramedic
* > 18 years
* < 60 years

Exclusion Criteria:

* pregnant
* lay rescuers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The average achieved cardiac output | after 10 minutes
  The main goal of the study is the average achieved cardiac output. Data acquisition is carried out on a resuscitation-manikin which can measure compression-rate (CR) and compression-depth (CD). The data are recorded by a computer during the CPR. To calculate the cardiac output, we multiply the average CR [1/min] with the average CD [mm] during the 10 min manikin-resuscitation. The thus obtained average cardiac-output (CO = CR x CD), measured in [mm/min], will be compared in each group.

SECONDARY OUTCOMES:
Now-flow-time | after 10 minutes
  Second objective of the study is the time without chest-compression during the 10 minutes ALS-CPR. The now-flow-time is read out of the recorded manikin-data specify, in [min] and [sec]. As a result, the average now-flow-time in each group will be calculated and compared for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Braunecker, MD, Principal Investigator — University Hospital Cologne; Jochen Hinkelbein, MD, Principal Investigator — University Hospital Cologne; Jan Hilgers, MD, Principal Investigator — University Hospital Cologne
Locations (1):
- Uniklinik Köln, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Schmitz J, Ernst C, Varghese LJK, Kerkhoff S, Jansen G, Hinkelbein J. A two-rescuer-method significantly alters CPR-quality during cardiopulmonary resuscitation in an airliner cabin - a randomized, controlled manikin trial. Sci Rep. 2025 Dec 10;15(1):43585. doi: 10.1038/s41598-025-30996-1. PMID 41372341